CLINICAL TRIAL: NCT03526549
Title: A Phase 3b, Open-Label, Long-Term Study to Evaluate the Safety and Temporal Pattern of Response of EN3835 in the Treatment of Edematous Fibrosclerotic Panniculopathy
Brief Title: Long-Term Study of EN3835 (CCH-aaes) in Edematous Fibrosclerotic Panniculopathy (Cellulite)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-304
Record Dates: First submitted 2018-04-25; First posted 2018-05-16 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite
MeSH Terms: conditions — Cellulite | interventions — Observation

STUDY DESIGN:
Masking Description: Investigators, participants, and site personnel were blinded to the treatment administered in the EN3835-302/303 parent studies until all Day 180 visit assessments were completed.
  CCH-aaes retreatment in this study was provided in an open-label manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CCH-aaes Treatment in Parent Studies (EN3835-302/303) (Experimental): Participants who received CCH-aaes treatment in EN3835-302/303 were followed for 180 days of observation with no treatment. Participants who were identified as received CCH-aaes in the parent studies following the 180-day Observation Phase and entered the Open-label Phase of the study. Participants in the Open-label Phase who qualified for, and opted for, retreatment were administered CCH-aaes up to 1.68 mg at 3 treatment sessions, at 21-day intervals.
  Interventions: Biological: CCH-aaes; Other: Observation
- Placebo Treatment in Parent Studies (EN3835-302/303) (Other): Participants who received placebo in the parent studies, were followed for 180 days of observation with no treatment. After Day 180, all participants who received placebo during the double-blind parent studies were discontinued. No treatment was administered.
  Interventions: Other: Observation

INTERVENTIONS:
Biological: CCH-aaes — Administered to participants who qualified for, and opted for, retreatment.
  Other Names: EN3835; QWO™
  Arms: CCH-aaes Treatment in Parent Studies (EN3835-302/303)
Other: Observation — No treatment administered during 180 days of observation.

SUMMARY:
A Phase 3b, Open-Label Extension Study to evaluate safety and how long response of EN3835 (Collagenase Clostridium Histolyticum [CCH]-aaes) lasts in the treatment of Cellulite.

DETAILED DESCRIPTION:
This study included participants who completed EN3835-302 (NCT03428750) or EN3835-303 (NCT03446781) double-blind parent studies. The first part of this study consisted of an observational period conducted in a blinded fashion and where no treatments were administered between Day 71 of the parent studies and Day 180 in this Open-label extension study. Once these participants were unblinded at Day 180, only participants who received active CCH-aaes in the parent studies remained in this study and those who received placebo in the parent studies were not eligible to continue in the Open-label study. Assessments made at the Day 71/(End of Study [EOS]) visit of the parent studies served as initial screening assessments for this study.

In the Open-label Phase of the study, all participants who qualified for, and opted for, retreatment were administered CCH-aaes at 3 treatment sessions at 21-day intervals.

ELIGIBILITY:
Key Inclusion Criteria

All Participants (Through Day 180):

1. Voluntarily sign and date an informed consent agreement
2. Have participated in and completed the double-blind Phase 3 study EN3835-302 or EN3835-303
3. Be willing to apply sunscreen to the buttocks before each exposure to the sun and/or tanning booths while participating in the study
4. Be judged to be in good health
5. Be willing and able to cooperate with the requirements of the study
6. Be able to read, complete and understand the participant reported outcomes rating instruments in English.

Key Inclusion Criteria for Participants Eligible for Retreatment:

1. Have a negative pregnancy test and using a stable and effective contraception method.

Key Exclusion Criteria

All Participants (Through Day 180):

1. Intends to or has used any of the local applications/therapies/injections/procedures that restricts study participation
2. Intends to use tanning spray or tanning booths during this period
3. Has received or intends to receive an investigational drug or treatment, other than the treatment received in study EN3835-302/303 during this period
4. Any other condition(s) that, in the Investigator's opinion, might indicate the participant to be unsuitable for the study

Additional Exclusion Criteria may apply Post Day 180:

1. Has received any collagenase treatments at any time since completion of the double-blind study (EN3835-302 or EN3835-303).

Key Exclusion Criteria for Participants Eligible for Retreatment:

1. Has systemic conditions (coagulation disorders, malignancy, keloidal scar, abnormal wound healing) that restricts study participation

* Has local (in areas to be treated) conditions (thrombosis, vascular disorder, active infection/inflammation, skin laxity, flaccidity and/or skin sagging, active cutaneous alteration, tattoo/mole) that restricts study participation
* Requires anticoagulant or antiplatelet medication during the study
* Prior to and during the course of retreatment, is nursing or providing breast milk in any manner, intends to become pregnant during the study, or intends to use tanning spray or tanning booths during the study
* Has received an investigational drug or treatment, other than treatment in study EN3835-302/303, within 30 days before retreatment with study drug
* Has a known systemic allergy to collagenase or any other excipient of study drug
* Has received any collagenase treatments at any time since completion of the double-blind study
* Any other condition(s) that, in the Investigator's opinion, might indicate the participant to be unsuitable for retreatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chajko, Study Director — Endo Pharmaceuticals
Locations (42):
- United States (42):
  - Endo Clinical Trial Site #3, Glendale, Arizona
  - Endo Clinical Trial Site #11, Scottsdale, Arizona
  - Endo Clinical Trial Site #41, North Little Rock, Arkansas
  - Endo Clinical Trial Site #14, Encinitas, California
  - Endo Clinical Trial Site #9, Long Beach, California
  - Endo Clinical Trial Site #35, Murrieta, California
  - Endo Clinical Trial Site #42, Newport Beach, California
  - Endo Clinical Trial Site #17, Oceanside, California
  - Endo Clinical Trial Site #39, San Diego, California
  - Endo Clinical Trial Site #23, Greenwood Village, Colorado
  - Endo Clinical Trial Site #38, Boca Raton, Florida
  - Endo Clinical Trial Site #8, Coral Gables, Florida
  - Endo Clinical Trial Site #40, Largo, Florida
  - Endo Clinical Trial Site #27, Miami, Florida
  - Endo Clinical Trial Site #36, Miami, Florida
  - Endo Clinical Trial Site #20, Snellville, Georgia
  - Endo Clinical Trial Site #19, Meridian, Idaho
  - Endo Clinical Trial Site #34, Chicago, Illinois
  - Endo Clinical Trial Site #30, Indianapolis, Indiana
  - Endo Clinical Trial Site #16, Metairie, Louisiana
  - Endo Clinical Trial Site #10, New Orleans, Louisiana
  - Endo Clinical Trial Site #25, New Orleans, Louisiana
  - Endo Clinical Trial Site #33, Quincy, Massachusetts
  - Endo Clinical Trial Site #18, Washington, Missouri
  - Endo Clinical Trial Site #4, Omaha, Nebraska
  - Endo Clinical Trial Site #24, Mount Kisco, New York
  - Endo Clinical Trial Site #32, New York, New York
  - Endo Clinical Trial Site #12, New York, New York
  - Endo Clinical Trial Site #15, New York, New York
  - Endo Clinical Trial Site #29, New York, New York
  - Endo Clinical Trial Site #26, Cincinnati, Ohio
  - Endo Clinical Trial Site #5, Nashville, Tennessee
  - Endo Clinical Trial Site #22, Austin, Texas
  - Endo Clinical Trial Site #6, Beaumont, Texas
  - Endo Clinical Trial Site #13, Houston, Texas
  - Endo Clinical Trial Site #7, Houston, Texas
  - Endo Clinical Trial Site #28, Pflugerville, Texas
  - Endo Clinical Trial Site #21, San Antonio, Texas
  - Endo Clinical Trial Site #37, Sugar Land, Texas
  - Endo Clinical Trial Site #31, Salt Lake City, Utah
  - Endo Clinical Trial Site #1, Charlottesville, Virginia
  - Endo Clinical Trial Site #2, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Rollover participants from the parent studies, EN3835-302 or EN3835-303 (CCH-aaes-treated or placebo-treated) were unblinded at Day 180 (after observation phase) and only participants who received active CCH-aaes remained in this Open-label Phase of the study.
Groups:
- CCH-aaes Treatment in Parent Studies EN3835-302/303: Participants who received CCH-aaes treatment in the parent studies were followed for 180 days of observation with no treatment. Participants who were identified as received CCH-aaes in the parent studies following the 180-day Observation Phase entered the Open-label Phase. Participants in the Open-label Phase who qualified for, and opted for, retreatment were administered CCH-aaes up to 1.68 mg at 3 treatment sessions, at 21-day intervals.
- Placebo Treatment in Parent Studies EN3835-302/303: Participants who received placebo in the parent studies, were followed for 180 days of observation with no treatment. After Day 180, all participants who received placebo during the double-blind parent studies were discontinued.
Period: 180 Days Observational Phase
Arm/Group | CCH-aaes Treatment in Parent Studies EN3835-302/303 | Placebo Treatment in Parent Studies EN3835-302/303
Started | 243 | 240
Completed Day 180 | 243 | 240
Completed (Completed 180 days of observation and consented to continue in the Open-label Phase.) | 202 | 0 (After Day 180, all participants who received placebo during the double-blind studies were discontinued.)
Not Completed | 41 | 240
Not completed — Participants who Received Placebo in Parent Studies were Discontinued | 0 | 238
Not completed — Withdrawal by Subject | 40 | 2
Not completed — Lost to Follow-up | 1 | 0
Period: Open-label Phase
Arm/Group | CCH-aaes Treatment in Parent Studies EN3835-302/303 | Placebo Treatment in Parent Studies EN3835-302/303
Started | 202 (All participants who received CCH-aaes in parent studies and consented to continue in the Open-label Phase of the study.) | 0
CCH-aaes Retreatment (Participants who qualified and opted for CCH-aaes retreatment in the Open-label Phase.) | 55 | 0
Completed | 104 | 0
Not Completed | 98 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 54 | 0
Not completed — Lost to Follow-up | 35 | 0
Not completed — Other than Specified | 5 | 0

BASELINE CHARACTERISTICS:
Population: Day 180 Observation Phase Population: All rollover participants who completed the parent studies (EN3835-302 or EN3835-303) (CCH-aaes-treated or placebo-treated).
Groups:
- Overall Participants: Participants who received CCH-aaes or placebo treatment in the parent studies were followed for 180 days of observation with no treatment. Participants who were identified as received CCH-aaes in the parent studies following the 180-day Observation Phase entered the Open-label Phase. Participants in the Open-label Phase who qualified for, and opted for, retreatment were administered CCH-aaes up to 1.68 mg at 3 treatment sessions, at 21-day intervals and participants who received placebo during the parent studies were discontinued.
Arm/Group | Overall Participants
Number analyzed (Participants) | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 483
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : American Indian or Alaska Native | 2
  Race : Asian | 3
  Race : Black or African American | 87
  Race : Native Hawaiian or Other Pacific Islander | 1
  Race : White | 382
  Race : Other | 2
  Race : Multiple | 6
  Ethnicity: Hispanic or Latino | 90
  Ethnicity: Not Hispanic or Latino | 393
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.00 (7.108)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any unfavorable or unintended change in body structure (signs), body function (symptoms), laboratory result, or worsening of a pre-existing condition associated temporally with the use of the study medication whether or not considered related to the study medication. TEAEs were defined as any AEs with a start date equal to or after the date of the first injection. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to Day 1080
Population: Day 180 Observation Phase Population included all rollover participants who completed the parent studies (EN3835-302 or EN3835-303) (CCH-aaes-treated or placebo-treated). Open-label Phase Population included participants who received CCH-aaes in the parent study and who consented to continue in the Open-label Phase of the study. Open-label CCH-aaes Retreatment Population included participants in the Open-label Phase who qualified for, and opted for, retreatment with CCH-aaes.
Measure: Count of Participants; unit: Participants
Groups:
- Day 180 Observation Phase: CCH-aaes Treatment in Parent Studies EN3835-302/303: Participants who received CCH-aaes in the parent studies, were followed for 180 days of observation with no treatment.
- Day 180 Observation Phase: Placebo Treatment in Parent Studies EN3835-302/303: Participants who received placebo in the parent studies, were followed for 180 days of observation with no treatment.
- Open-label Phase (Prior to Retreatment): Participants who were identified as received CCH-aaes in the parent studies following the 180-day Observation Phase and who consented to continue in the Open-label Phase of the study.
- Open-label CCH-aaes Retreatment Phase: Participants in the Open-label Phase who qualified for, and opted for, retreatment were administered CCH-aaes up to 1.68 mg at 3 treatment sessions, at 21-day intervals.
Arm/Group | Day 180 Observation Phase: CCH-aaes Treatment in Parent Studies EN3835-302/303 | Day 180 Observation Phase: Placebo Treatment in Parent Studies EN3835-302/303 | Open-label Phase (Prior to Retreatment) | Open-label CCH-aaes Retreatment Phase
Number analyzed (Participants) | 243 | 240 | 202 | 55
Participants | 58 | 29 | 43 | 45

2. Primary Outcome: Percentage of Participants Who Were Seropositive for Anti-Drug Antibodies (ADAs) After CCH-aaes Treatment
Description: Serum samples were analyzed for ADAs. The percentage of participants who developed ADAs (seropositive results) during the Open-label Phase of the study are reported.
Time Frame: From Day 180 (Open-label Phase) up to Day 1080
Population: Open-label Phase Population included participants who received CCH-aaes in the parent study and who consented to continue in the Open-label Phase of the study. Open-label CCH-aaes Retreatment Population included participants in the Open-label Phase who qualified for, and opted for, retreatment with CCH-aaes. Participants who received placebo during the parent studies did not continue in the Open-label Phase.
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Phase (Prior to Retreatment) | Open-label CCH-aaes Retreatment Phase
Number analyzed (Participants) | 202 | 55
percentage of participants | 98.2 | 100

3. Secondary Outcome: Time to 2-Level Reduction of Response in Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient Reported Photonumeric Cellulite Severity Scale (PR-PCSS)
Description: CR-PCSS and PR-PCSS assess improvement in cellulite severity using a 5-level scale ranging from "0" (None) to "4" (Severe). Time to reduction of response (days) was defined as the number of days from Screening assessment of composite improvement in cellulite severity in PR-PCSS and CR-PCSS to the time at which a 2-level composite worsening of response was observed for the first time.
Time Frame: From Day 180 (Open-label Observation Phase) up to Day 1080
Population: Participants who were treated with CCH-aaes and had a 2-level composite response in CR-PCSS and PR-PCSS in the parent studies and who consented to continue in the Open-label Phase of this study. Participants who had a 2-level reduction in response in CR-PCSS and PR-PCSS were to be assessed for time to event.
Measure: Number; unit: days
Arm/Group | Open-label Phase (Prior to Retreatment)
Number analyzed (Participants) | 20
days | NA — No participants had a 2-level reduction in response so it was not possible to calculate a time to a 2-level reduction in response.

4. Secondary Outcome: Time to 1-Level Reduction of Response in CR-PCSS and PR-PCSS
Description: CR-PCSS and PR-PCSS assess improvement in cellulite severity using a 5-level scale ranging from "0" (None) to "4" (Severe). Time to reduction of response (days) was defined as the number of days from Screening assessment of composite improvement in cellulite severity in CR-PCSS and PR-PCSS to the time at which 1-level composite worsening of response was observed for the first time.
Time Frame: From Day 180 (Open-label Observation Phase) up to Day 1080
Population: This assessment includes both 1-level and 2-level composite responders in the parent studies who had a 1-level reduction of response in CR-PCSS and PR-PCSS.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Open-label Phase (Prior to Retreatment)
Number analyzed (Participants) | 24
days | 356.5 (232.43)

5. Secondary Outcome: Time to Complete Loss of Response in CR-PCSS and PR-PCSS
Description: CR-PCSS and PR-PCSS assess improvement in cellulite severity using a 5-level scale ranging from "0" (None) to "4" (Severe). Complete loss of response is defined as both CR-PCSS and PR-PCSS ratings returned to the baseline severity of the double-blind study or worse for both the buttocks. Time to complete loss of response (days) was defined as the number of days from Screening assessment of composite improvement in cellulite severity in CR-PCSS and PR-PCSS to the time at which complete loss of response was observed for the first time.
Time Frame: From Day 180 (Open-label Observation Phase) up to Day 1080
Population: This assessment includes both 1-level and 2-level composite responders in the parent studies who had complete loss of response in CR-PCSS and PR-PCSS.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Open-label Phase (Prior to Retreatment)
Number analyzed (Participants) | 6
days | 238.2 (85.75)

ADVERSE EVENTS:
Time Frame: Up to Day 1080
Description: Day 180 Observation Phase Population included all rollover participants who completed the parent studies (CCH-aaes-treated or placebo-treated). Open-label Phase Population included participants who received CCH-aaes in the parent study and who consented to continue in the Open-label Phase of the study. Open-label CCH-aaes Retreatment Population included participants in the Open-label Phase who qualified for, and opted for, retreatment with CCH-aaes.
Groups:
- Day 180 Observation Phase: CCH-aaes Treatment in Parent Studies EN3835-302/303: Participants who received CCH-aaes in the parent studies were followed for 180 days of observation with no treatment.
- Day 180 Observation Phase: Placebo Treatment in Parent Studies EN3835-302/303: Participants who received placebo in the parent studies were followed for 180 days of observation with no treatment.
Arm/Group | Day 180 Observation Phase: CCH-aaes Treatment in Parent Studies EN3835-302/303 | Day 180 Observation Phase: Placebo Treatment in Parent Studies EN3835-302/303 | Open-label Phase (Prior to Retreatment) | Open-label CCH-aaes Retreatment Phase
All-Cause Mortality (participants affected / at risk) | 0/243 | 0/240 | 0/202 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/243 | 1/240 | 3/202 | 3/55
Other Adverse Events (participants affected / at risk) | 27/243 | 0/240 | 7/202 | 31/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Day 180 Observation Phase: CCH-aaes Treatment in Parent Studies EN3835-302/303 (N=243) | Day 180 Observation Phase: Placebo Treatment in Parent Studies EN3835-302/303 (N=240) | Open-label Phase (Prior to Retreatment) (N=202) | Open-label CCH-aaes Retreatment Phase (N=55)
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Day 180 Observation Phase: CCH-aaes Treatment in Parent Studies EN3835-302/303 (N=243) | Day 180 Observation Phase: Placebo Treatment in Parent Studies EN3835-302/303 (N=240) | Open-label Phase (Prior to Retreatment) (N=202) | Open-label CCH-aaes Retreatment Phase (N=55)
Injection site bruising (General disorders) | 12 | 0 | 0 | 31
Injection site discolouration (General disorders) | 10 | 0 | 2 | 4
Corona virus infection (Infections and infestations) | 0 | 0 | 5 | 3
Injection site pain (General disorders) | 0 | 0 | 0 | 10
Injection site pruritus (General disorders) | 0 | 0 | 0 | 9
Injection site erythema (General disorders) | 0 | 0 | 0 | 6
Injection site nodule (General disorders) | 3 | 0 | 0 | 4
Injection site swelling (General disorders) | 1 | 0 | 0 | 4
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 3
Injection site induration (General disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03526549/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03526549/SAP_001.pdf